CLINICAL TRIAL: NCT06730997
Title: Clinicopathological Features of Renal Cell Carcinoma in Young Patients and it's Influence on the Survival Outcome
Brief Title: Clinicopathological Features of Renal Cell Carcinoma in Young Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Gamal Abdelaziz Farrag, physion, Assiut University
Other Study IDs: Renal cell carcinoma
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Clinicopathologic Characters of Renal Cell Carcinoma in Young Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Analysis of Clinicopathologic Characters of Renal Cell Carcinoma in Young Patients and their influence on the survival outcomes

DETAILED DESCRIPTION:
Worldwide, RCC accounts for 2-3% of All adult malignancies and the 8th most commonly diagnosed primary cancer among all adults.

Representing 3rd place among urinary system tumors. Most of RCC occurs in old age while about 7% occurs in younger adults below 40 years.

Recently the published data about the tumor Clinco-pathological features, treatment response and outcomes were different in young adults than older patients, where some data showed favorable features and survivals, while other showed negative ones.

ELIGIBILITY:
Inclusion Criteria:

* Age < 40 years

  * Patients proven to have RCC
  * Patients eligible to receive treatment

Exclusion Criteria:

* Second malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with renal cell carcinoma 40 years or younger at Radiation Oncology Department, South Egypt Cancer Institute, clinical oncology Assuit University at the period from 2015 to 2022
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of Clinicopathologic Characters of Renal Cell Carcinoma in Young Patients and their influence on the survival outcomes | Analysis of Clinicopathologic Characters of Renal Cell Carcinoma in Young Patient in period from 2010 -2024
  Analysis of Clinicopathologic Characters of Renal Cell Carcinoma in Young Patients and their influence on the survival outcomes

REFERENCES:
- [Background] Lipworth L, Tarone RE, McLaughlin JK. The epidemiology of renal cell carcinoma. J Urol. 2006 Dec;176(6 Pt 1):2353-8. doi: 10.1016/j.juro.2006.07.130. PMID 17085101
- [Background] Suh JH, Oak T, Ro JY, Truong LD, Ayala AG, Shen SS. Clinicopathologic features of renal cell carcinoma in young adults: a comparison study with renal cell carcinoma in older patients. Int J Clin Exp Pathol. 2009;2(5):489-93. Epub 2009 Jan 30. PMID 19294008
- [Background] Moch H, Cubilla AL, Humphrey PA, Reuter VE, Ulbright TM. The 2016 WHO Classification of Tumours of the Urinary System and Male Genital Organs-Part A: Renal, Penile, and Testicular Tumours. Eur Urol. 2016 Jul;70(1):93-105. doi: 10.1016/j.eururo.2016.02.029. Epub 2016 Feb 28. PMID 26935559